CLINICAL TRIAL: NCT03834974
Title: Using a Narrative-Based Approach to Reducing Indoor Tanning
Brief Title: Social Media Indoor Tanning Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H19-033; R21CA226133-01 (NIH)
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sun Safety Social Media Challenge (Experimental): During this 4-week intervention, participants will be incentivized to create sun safety social media messages that will be distributed on our sun safety Twitter and Facebook feeds.
  Interventions: Behavioral: Sun Safety Social Media Challenge
- Digital Health Social Media Challenge (Active Comparator): During this 4-week intervention, participants will be incentivized to create posts that promote the use of technology to engage in healthy lifestyle behaviors (diet, exercise) on our digital health Twitter and Facebook feeds.
  Interventions: Behavioral: Digital Health Social Media Challenge

INTERVENTIONS:
Behavioral: Sun Safety Social Media Challenge — Participants will attend a webinar to learn how to create effective social media posts about sun safety and be oriented to the social media accounts on which the messages will be posted. They will be informed that posts should include a sun safety message (e.g., promoting sunscreen use and protective clothing/hats or discouraging risk behaviors like tanning and burning). They will be encouraged to be creative so that the message gets likes and shares. Participants will be encouraged to follow the feeds to see the engagement on their posts, to share the posts in their feed, and to see other participants' posts. Participants will receive a $10 Amazon gift card per post for a maximum of 6 posts ($60). The participant who created the post that receives the most likes, comments, and shares each week will win a $50 Amazon gift card.
  Arms: Sun Safety Social Media Challenge
Behavioral: Digital Health Social Media Challenge — Participants will attend a webinar to learn how to create effective social media posts about using technology to get healthy and be oriented to the social media accounts on which the messages will be posted. They will be informed that posts should mention some way that technology (e.g., mobile apps, wearables) can be used to promote a healthy habit (e.g., diet, exercise). They will be encouraged to be creative so that the message gets likes and shares. Participants will be encouraged to follow the feeds to see the engagement on their posts, to share the posts in their feed, and to see other participants' posts. Participants will receive a $10 Amazon gift card per post for a maximum of 6 posts ($60). The participant who created the post that receives the most likes, comments, and shares each week will win a $50 Amazon gift card.
  Arms: Digital Health Social Media Challenge

SUMMARY:
The purpose of this research is to develop a social media delivered intervention to reduce unprotected sun exposure in young adults with a history of tanning.

DETAILED DESCRIPTION:
We will use social marketing theory and a user-centered design approach to develop a social media intervention that engages young adults with a history of tanning to practice sun safety behaviors. We will incentivize young adults who have a history of tanning to create social media posts that encourage their peers to engage in sun safety. Focus groups of tanners guided the development of the intervention. Investigators will conduct a pilot feasibility trial where participants will be randomized to a condition in which they are incentivized to create sun safety social media messages to be posted on a sun safety social media account or a condition in which they are incentivized to create social media messages about how to use technology to support healthy lifestyle behaviors to be posted on a health technology social media account. The intervention will last 4 weeks. Feasibility outcomes include recruitment, retention, acceptability, participation, social media message engagement (likes, comments, shares), persuasive impact of messages, unprotected sun exposure, sun protection, and tanning behavior. This work will inform a fully powered randomized trial testing the efficacy of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30
* Tanned indoors or outdoors at least once in the past year
* Intends to tan indoors or outdoors this summer
* Daily user of any social media platform

Exclusion Criteria:

* No smartphone
* Does not use a social media platform daily
* Lives in a state with an average temperature <75 degrees in May
* Inability to provide consent due to mental illness or a cognitive impairment
* Non-English speaking
* Prisoner

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry L Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Pagoto SL, Waring ME, Groshon LC, Rosen AO, Schroeder MW, Goetz JM. Proof-of-Concept Feasibility Trial of a Dissonance-Based Sun Safety Intervention for Young Adult Tanners. Ann Behav Med. 2022 Aug 2;56(8):830-841. doi: 10.1093/abm/kaab116. PMID 35179176

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24.0 [20.0 to 28.0] | 23.5 [20.5 to 27.5] | 24.0 [20.0 to 28.0]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Number of participants belonging to each gender
  Participants
    Gender: Female | 28 | 27 | 55
    Gender: Male | 5 | 5 | 10
    Gender: Non-Binary/Third Gender | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Number of participants belonging to each race/ethnicity
  Participants
    Race/ethnicity: Non-Hispanic White | 18 | 17 | 35
    Race/ethnicity: Non-Hispanic Black/African American | 1 | 1 | 2
    Race/ethnicity: Hispanic/Latino of any race | 5 | 7 | 12
    Race/ethnicity: Non-Hispanic Asian | 9 | 3 | 12
    Race/ethnicity: Native Hawaiian or Other Pacific Islander, Native, Other, and Multiracial (Non-Hispanic) | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: The number of completed respondents to recruitment ads, number of respondents eligible at initial screening, and number of respondents who completed baseline.
Time Frame: Baseline
Population: All prospective participants
Measure: Count of Participants; unit: Participants
Groups:
- Prospective Participants: All prospective participants
Arm/Group | Prospective Participants
Number analyzed (Participants) | 549
Participants
  Number of completed respondents to recruitment ads | 549
  Number of respondents eligible at initial screening | 79
  Number of respondents who completed baseline | 66

2. Primary Outcome: Retention
Description: The % of participants in each condition who complete the follow-up assessment.
Time Frame: 4-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants | 34 | 32

3. Primary Outcome: Acceptability
Description: Number of participants who selected agree or strongly agree on 5-point Likert scale rating of how likely participants would be to recommend the intervention to a friend, and how likely they would be to participate again.
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants
  I would participate in this study competition on this health topic again. | 31 | 29
  I would recommend this study competition to a friend. | 32 | 31

4. Primary Outcome: Participation
Description: The number of posts created by participants
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Number; unit: number of posts
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
number of posts | 148 | 129

5. Primary Outcome: Post Engagement
Description: The median number of likes, shares and retweets, and unique commenters each participant post received.
Time Frame: 4 weeks
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: Engagement
Units Other Than Participants: Posts
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Number analyzed (Posts) | 148 | 129
Engagement
  Twitter Likes and Facebook Reactions | 4 [2 to 8] | 2 [1 to 7]
  Twitter Retweets and Facebook Shares | 2 [1 to 5] | 0 [0 to 3]
  Unique Commenters on Facebook and Twitter | 0 [0 to 2] | 0 [0 to 2]

6. Primary Outcome: Desirability of Tanning
Description: Scale measuring participants' belief that a tan is attractive. Scale ranges from 0-12 with higher scores indicating higher levels of belief that a tan is attractive.
Time Frame: Baseline
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
score on a scale | 11 [9 to 12] | 11 [9 to 12]

7. Primary Outcome: Desirability of Tanning
Description: as for outcome 6
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
score on a scale | 10 [9 to 12] | 10.5 [9 to 12]

8. Primary Outcome: Desirability of Tanning Alternatives
Description: Average score on items relating to tanning alternative desirability. Scale ranges from 1 to 5, with higher scores indicating more positive attitudes towards tanning alternatives.
Time Frame: Baseline
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
score on a scale | 3.0 (1.2) | 3.5 (1.2)

9. Primary Outcome: Desirability of Tanning Alternatives
Description: as for outcome 8
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
score on a scale | 2.8 (1.1) | 3.5 (1.1)

10. Primary Outcome: Persuasive Impact of Participant Messages
Description: The mean of participants ratings for how persuasive they found each post (other than those they created) on a scale of 0-100, with higher scores indicating more persuasive.
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: score on a sliding scale
Units Other Than Participants: Posts
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Number analyzed (Posts) | 148 | 129
score on a sliding scale | 62.2 (13.3) | 62.5 (14.7)

11. Primary Outcome: Contamination
Description: The number of participants who report they saw the opposite conditions Facebook or Twitter feeds.
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants | 7 | 10

12. Secondary Outcome: Outdoor Tanning Intentions
Description: Three items assessed intentions to tan even once, intentions to tan regularly in the next year, and intentions to quit on a 7-point scale (0=definitely will not, 6=definitely will).
Time Frame: Baseline
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
score on a scale
  Tan outside in the sun sometime later in my life. | 6.0 [4.0 to 6.0] | 6.0 [5.0 to 6.0]
  Tan outside in the sun more than 10 times in the next year. | 6.0 [3.0 to 6.0] | 6.0 [3.0 to 6.0]
  Quit tanning outside in the next year. | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 1.0]

13. Secondary Outcome: Outdoor Tanning Intentions
Description: as for outcome 12
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
score on a scale
  Tan outside in the sun sometime later in my life. | 5.0 [3.0 to 6.0] | 6.0 [5.0 to 6.0]
  Tan outside in the sun more than 10 times in the next year. | 3.0 [1.0 to 4.0] | 5.0 [3.0 to 6.0]
  Quite tanning outside in the next year. | 1.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
Statistical Analysis 1: Comparison: Sun Safety Social Media Challenge vs Digital Health Social Media Challenge; Null hypothesis: There would be no difference in change in intent to tan outdoors 10 or more times in the next year; Test type: Superiority; p < 0.0286, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Sun Safety Social Media Challenge vs Digital Health Social Media Challenge; Null hypothesis: There would be no difference in change in in intent to tan later in life; Test type: Superiority; p = 0.0937, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Sun Exposure
Description: How many hours the participant spent outside per week between the hours of 10am and 4pm.
Time Frame: Baseline
Population: all randomized participants
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
hours per week | 16.1 (10.4) | 15.6 (7.3)

15. Secondary Outcome: Sun Exposure
Description: How many hours the participant spent outside per week between 10am and 4pm
Time Frame: 4-week follow-up
Population: all randomized participants
Measure: Mean (Standard Deviation); unit: hours per week
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
hours per week | 11.4 (5.9) | 13.2 (8.2)

16. Secondary Outcome: Outdoor Tanning
Description: How many times in the last 4 weeks the participant went outside for the purpose of tanning in the sun.
Time Frame: Baseline
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: outdoor tanning sessions
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
outdoor tanning sessions | 4.0 [0.0 to 8.0] | 5.0 [2.0 to 10.0]

17. Secondary Outcome: Outdoor Tanning
Description: How many times in the last 4 weeks the participant went outside for the purpose of tanning in the sun.
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: outdoor tanning sessions
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
outdoor tanning sessions | 0.0 [0.0 to 1.0] | 2.0 [0.5 to 5.0]
Statistical Analysis 1: Comparison: Sun Safety Social Media Challenge vs Digital Health Social Media Challenge; Null hypothesis: There would be no difference in tanning outside at follow-up; Test type: Superiority; p < 0.0002, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Sun Protection
Description: Number of participants who reported using sun protection (sunscreen, protective clothing) often or always in the past month
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants
  How often did you wear sunscreen? | 18 | 16
  How often did you wear a shirt with sleeves that covered your shoulders? | 15 | 9
  How often did you wear a hat? | 8 | 2
  How often did you stay in the shade or under an umbrella? | 3 | 0
  How often did you wear sunglasses? | 19 | 21

19. Secondary Outcome: Sun Protection
Description: as for outcome 18
Time Frame: 4-week follow-up
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants
  How often did you wear sunscreen? | 19 | 16
  How often did you wear a shirt with sleeves that covered your shoulders? | 20 | 14
  How often did you wear a hat? | 6 | 4
  How often did you stay in the shade or under an umbrella? | 12 | 5
  How often did you wear sunglasses? | 18 | 22

20. Secondary Outcome: Indoor Tanning Behavior
Description: Number of indoor tanning visits in the previous month
Time Frame: Baseline
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: indoor tanning sessions
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
indoor tanning sessions | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]

21. Secondary Outcome: Indoor Tanning Behavior
Description: Number of indoor tanning visits in the previous month
Time Frame: 4 weeks
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: indoor tanning sessions
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
indoor tanning sessions | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

22. Secondary Outcome: Sunburn
Description: Number of participants with 1 or more sunburns in the past month
Time Frame: baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants | 15 | 13

23. Secondary Outcome: Sunburn
Description: Number of participants with 1 or more sunburns in the past month
Time Frame: 4 weeks
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 34 | 32
Participants | 5 | 2

24. Secondary Outcome: Outdoor Tanning Duration
Description: Median reported average number of minutes tanned per episode in the past 4 weeks, among participants who tanned in the past 4 weeks.
Time Frame: 4 weeks
Population: Randomized participants who reported tanning one or more times in the past 4 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 10 | 24
minutes | 45.0 [25.0 to 120.0] | 60.0 [30.0 to 72.5]

25. Secondary Outcome: Outdoor Tanning Duration
Description: as for outcome 24
Time Frame: Baseline
Population: Randomized participants who reported tanning one or more times in the past 4 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
Number analyzed (Participants) | 24 | 25
minutes | 60.0 [42.5 to 105.0] | 60.0 [45.0 to 120.0]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Sun Safety Social Media Challenge | Digital Health Social Media Challenge
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03834974/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03834974/SAP_001.pdf
  • Informed Consent Form (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03834974/ICF_002.pdf